CLINICAL TRIAL: NCT02590653
Title: Assessment of the Effects of Aggressive Atorvastatin Therapy on Myocardial Deformation Characteristics, Vascular Rigidity, 24 Hour ECG Monitoring Parameters and Quality of Life in Patients With STEMI
Brief Title: Assessment of the Effects of Atorvastatin Therapy on Myocardial Deformation Characteristics, in Patients With STEMI
Acronym: CONTRAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penza State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSU/T-253
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Myocardial Infarction
Keywords: STEMI; myocardial strain; atorvastatin
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Group A patients will start atorvastatin at a dose of 80 mg/day between 24 and 96 hours after the onset of STEMI
  Interventions: Drug: Atorvastatin
- Group K (Active Comparator): Group K patients will start atorvastatin at a dose of 20 mg/day between 24 and 96 hours after the onset of STEMI
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Lipid-lowering therapy
  Other Names: Statin

SUMMARY:
The primary goal

• To assess the effect of atorvastatin in patients treated since the first 24-96 hours of the disease on the parameters of global and regional myocardial deformation in the infarcted area and the structural and functional properties of arteries at day 7, at 12, 24, 36 and 48 weeks of treatment;

The secondary goals. To evaluate the effect of treatment:

* on the parameters of the global and regional myocardial deformation in the intact area on day 7, on 12, 24, 36 and 48 weeks of treatment;
* on the parameters of the global and regional myocardial deformation depending on the degree of coronary blood flow restoration by thrombolysis in myocardial infarction (TIMI)
* on systolic and diastolic left ventricular function in the presence of initial impairments, or absence of the negative dynamics of these parameters in case of normal baseline values;
* on the clinical diagnostic criteria for the development or progression of heart failure;
* the dynamics of the duration and extent of myocardial ischemia according to the daily ECG monitoring on day 7, at 12, 24, 36 and 48 weeks of treatment;
* the appearance of new prognostically significant cardiac arrhythmias
* on the pulse wave velocity
* the thickness of the intima-media complex (IMT); 200 patients are planned to be include in a randomized, single-center, open, prospective, controlled clinical trial, the enrollment will be held at the Department of "Therapy" of Medical Institute of Penza State University.

Definition of the study group:

The patients with STEMI (myocardial infarction with ST-segment elevation) will be included in the study

* Group 1 STEMI - 100 patients receiving atorvastatin 80 mg / day for 48 weeks;
* Group 2 STEMI - 100 patients receiving atorvastatin 20 mg / day for 48 weeks Planned number of patients: Pre-Screening - 300 subjects; screening and randomization - 200 subjects.

Patients will be randomized by random number generation to include in the group 1 or 2. All included patients will be on the standard basis therapy of the coronary artery disease, according to the national recommendation.

DETAILED DESCRIPTION:
1. Hypotheses:

1. Atorvastatin therapy directly results in improved deformation characteristics of hibernating myocardium due to its pleiotropic effects on endothelial dysfunction and atherosclerotic plaque stability, as well as stimulation of angiogenesis in ischemic zones of myocardium.
2. Long-term atorvastatin therapy improves the morphofunctional properties of large arteries and decreases the severity of endothelial dysfunction in patients with a history of myocardial infarction.
3. Atorvastatin causes an anti-ischemic effect, if used for a long time. 2.1. Primary objective To evaluate the effect of atorvastatin, when started between 24 and 96 hours after disease onset, on the parameters of global and regional myocardial deformation in the zone of infarction, as well as morphofunctional properties of arteries, on Day 7 and Weeks 12, 24, 36 and 48 of the treatment; 2.2. Secondary objectives. To evaluate:

   * the effect of treatment on the parameters of global and regional myocardial deformation in the zone of intact myocardium on Day 7 and Weeks 12, 24, 36 and 48 of the treatment;
   * the effect of treatment on the parameters of global and regional myocardial deformation depending on TIMI blood flow grade;
   * the effect of treatment on systolic and diastolic function of the left ventricle in patients with impaired left ventricular function at baseline, as well as the ability of this treatment to prevent deterioration of left ventricular function in patients with normal left ventricular function at baseline;
   * the effect of treatment on heart failure development and progression as assessed using the corresponding clinical diagnostic criteria;
   * the effect of treatment on duration and time course of myocardial ischemia using 24 hour ECG monitoring on Day 7 and Weeks 12, 24, 36 and 48 of treatment;
   * the effect of treatment on the appearance of new prognostically significant disorders of cardiac rhythm;
   * the effect of treatment on pulse wave velocity and cardio-ankle vascular index (CAVI);
   * the effect of treatment on intima-media thickness (IMT);
   * the effect of treatment on the results of automated quantitative vascular elasticity measurements, pulse wave and pulse pressure;
   * the effect of treatment on endothelial function using the reactive hyperemia test;
   * the effect of treatment on the time course of blood chemistry parameters (i.e., total cholesterol, HDL, LDL, triglycerides, creatinine, C-reactive protein (CRP), alanine transaminase (ALT), aspartate transaminase (AST) and creatinkinase (CK);
   * the safety of treatment;
   * the effect of treatment on patient's well-being and quality of life;
   * patient compliance with the therapy. 2.3. Scientific novelty of the study It is planned to study, for the first time, the effect of long-term aggressive statin therapy on the functional status of myocardium in the zone of ischemia, lesion and necrosis in patients with STEMI using the two-dimensional strain procedure.

It is planned, for the first time, to comprehensively study the effect of aggressive statin therapy on the status of vasculature, with measuring multiple parameters characterizing the morphofunctional status of elastic and muscular arteries in patients with documented coronary heart disease (CHD).

2.4. Clinical significance of study results. If the proposed hypotheses are confirmed after the primary endpoints described in Section 3 have been reached, new convincing evidence supporting the use of long-term aggressive treatment with Atorvastatin starting from the early stages of myocardial infarction will be obtained. Obviously, the clinical benefits will include the improved prognosis and decreased risk of repeated vascular events. Favorable effects of this therapy on the morphofunctional status of arterial vasculature will play an important role in the treatment of these patients. Positive results of this study can form the basis for planning and conducting larger studies on pleiotropic effects of Atorvastatin in patients with a history of myocardial infarction.

3. Primary endpoints

1. Statistically significant differences in spatial and velocity parameters of myocardial deformation in the zone of previous STEMI as compared to controls.
2. Statistically significant differences in spatial and velocity parameters of myocardial deformation in the intact zone after STEMI as compared to controls.
3. Statistically significant differences in intima-media thickness (IMT) according to echo tracking data as compared to controls.
4. Statistically significant differences in carotid-femoral pulse wave velocity and CAVI as compared to controls.

4. Planning and conducting the study. It is planned to include 200 patients in this randomized, open-label, single-center, prospective, controlled clinical study; these patients will be recruited at the Department of Therapy of the Penza State University Medical Institute.

4.1. Allocation to study groups:

Patients with STEMI will be included in this study:

Group 1: 100 patients with STEMI to receive atorvastatin at a dose of 80 mg per day for 48 weeks; Group 2: 100 patients with STEMI to receive atorvastatin at a dose of 20 mg per day for 48 weeks.

4.2. Planned number of patients: Prescreening - 300 patients; screening and randomization - 200 patients.

4.3. Study design. Patients will be randomized using sealed envelopes numbered with increasing serial numbers from 1 to 200; each envelope will contain information about patient inclusion into Group 1 or Group 2. Information about treatment schedule and dosing regimen will be provided separately.

4.3.1. Treatment regimen, dose titration strategy and combination treatment principles Patients meeting the inclusion criteria and not meeting the exclusion criteria will be included in the study.

Group A patients will start the treatment between 24 and 96 hours after the onset of STEMI:

• Atorvastatin at a dose of 80 mg per day.

Group K patients will start the treatment between 24 and 96 hours after the onset of STEMI:

• Atorvastatin at a dose of 20 mg per day.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Patients having physical and mental ability to participate in the study
3. Patients of both sexes aged 35 to 65 years
4. Presence of documented ST-elevation myocardial infarction confirmed by ECG, as well as troponin I and CK-MB levels.
5. Presence of hemodynamically relevant stenosis of one artery (i.e., the infarct-related artery) confirmed by coronary angiography (CAG), with the occlusion of other arteries not exceeding 30%.

Exclusion Criteria:

1. A history of repeat or recurrent myocardial infarction;
2. A history of chronic heart failure (CHF) III-IV by New-York Heart Association (NYHA);
3. Presence of left ventricular hypertrophy confirmed by echocardiography;
4. QRS complex exceeding 1.0;
5. Ejection fraction less than 40%;
6. Presence of hemodynamically relevant stenosis exceeding 30% in several coronary arteries confirmed by CAG;
7. Type 1 diabetes mellitus;
8. Type 2 diabetes mellitus requiring pharmacotherapeutic correction with insulin;
9. Any severe concurrent disease;
10. A history of acute cerebrovascular accident (ACVA) within the 6 month period preceding the study;
11. Active hepatic disease or liver enzyme elevation of unclear etiology more than 3 times higher than the upper limit of normal;
12. Hepatic failure or bilirubin elevation more than 1.5 times higher than the upper limit of normal;
13. Uncontrolled arterial hypertension (AH), with systolic blood pressure (SBP) exceeding 180 mm Hg and diastolic blood pressure (DBP) exceeding 110 mm Hg;
14. A history of heart rhythm and/or cardiac conduction disorder;
15. Inborn and/or acquired heart defects;
16. A history of aortic aneurysm;
17. Current existence of severe anemia (Hb < 100 g/L);
18. Chronic renal disease (creatinine clearance < 30 mL/min);
19. Uncorrected thyroid dysfunction, with hyper- or hypothyroidism;
20. Intolerance of statins;
21. Alcohol abuse and drug use;
22. Participation in other clinical studies within the last two months.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 2 years
  Myocardial infarction, Unstable angina, Cardiac death

SECONDARY OUTCOMES:
Global myocardial strain in the zone of previous STEMI and in the intact zone after STEMI | 2 years
  two-dimensional strain
Global myocardial strain rate in the zone of previous STEMI and in the intact zone after STEMI | 2 years
  two-dimensional strain
Intima-media thickness of carotid artery | 2 years
  echo-tracking
Carotid-femoral pulse wave velocity | 2 years
  Applanation tonometry
Cardiac-ankle vascular index | 2 years
  Volume sphygmography

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Oleynikov, prof., Principal Investigator — Head of Therapy Department
Locations (1):
- Valentin Oleynikov, Penza, Russia